CLINICAL TRIAL: NCT02467894
Title: Group-based Chronic Kidney Disease Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Michal L. Melamed, Associate Professor Of Medicine & Epidemiology & Population Health, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-3117
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Adherence; Exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group-based Care (Experimental): Participants who are randomized to group-based care will attend monthly outpatient clinic visits as part of a group of 8-10 patients with CKD and hypertension.
  Interventions: Other: Group-based Care
- Usual Care (No Intervention): Participants who are randomized to usual care will see their provider on clinic days when there is no group meeting.

INTERVENTIONS:
Other: Group-based Care — There will be self-care activities, blood pressure measurements and other vitals, including discussion of specific topics initiated by the participants.
  Arms: Group-based Care

SUMMARY:
A two-group randomized clinical trial testing whether group-based care is feasible and will help improve blood pressure control in adult and adolescent patients with chronic kidney disease and hypertension.

DETAILED DESCRIPTION:
This two-group RCT will enroll 100 subjects, adolescents over or equal to 12 years of age, and men and women over age of 21, with stage 3-4 and 5 CKD from various causes including diabetes and hypertension. Patients will be recruited from the Montefiore Medical Center Nephrology. The primary aim will be to assess feasibility of the intervention.

Informed consent will be obtained on all subjects. All subjects with meet with one of the investigators who will verbally explain to them the purpose of the study and the alternatives.

Blood and 24 hr urine test will be collected to assess for sodium, phosphorus, and serum creatinine. These tests will be used for experimental purposes only and will be collected at enrollment and 6 months visit.

There will be two arms, an arm randomized to Group-based care attending monthly outpatient clinic visits as part of a group and the other to usual care who will see their provider once a month for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Age ≥12 years old
* Sufficient hearing, vision, and proficiency in English or Spanish to comprehend low- literacy printed educational materials and participate in group sessions (assessed by provider)
* Adult: (¬>21 years): Systolic blood pressure >140 at two clinic visits in the past year or >160 at one visit and Adolescent: (12-21 years) systolic blood pressure >95 percentile (based on sex and age) at 2 clinic visits in the past year
* For adults: Stage 3-5 CKD (eGFR<60 ml/min/1.73m2)
* For adolescents: evidence of kidney damage (albuminuria, congenital anomalies of the kidney or urinary tract) and hypertension
* Prescription for anti-hypertensive medication (in adults)
* Unwillingness to accept random assignment
* Unwillingness to provide informed consent

Exclusion Criteria:

* Transplanted organ
* Rapidly deteriorating kidney function with the expectation for initiation of dialysis in less than 6 months
* Plans to relocate out of New York City in the next 6 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure control | 6 months
  The primary outcome will be blood pressure control (mean SBP <140 mmHg) as measured by 24-hour ambulatory blood pressure monitor.

OTHER OUTCOMES:
Accelerometer | 6 months
  Evaluate effects of group-based care on physical activity
Medication Adherence | 6 months
  Measured by the Morisky 8-item Medication Adherence scale.
Quality of Life | 6 months
  We will collect quality of life measurements using the Peds QL in the adolescent group and the SF-36 in the adult sample. We want to evaluate whether group-based care may lead to improved or worse reported quality of life in participants.
Health Resources and Services Administration (HRSA) | 6 months
  Evaluate patient and provider satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Johns TS, Brown DD, Litwin AH, Goldson G, Buttar RS, Kreimerman J, Lo Y, Reidy KJ, Bauman L, Kaskel F, Melamed ML. Group-Based Care in Adults and Adolescents With Hypertension and CKD: A Feasibility Study. Kidney Med. 2020 Apr 18;2(3):317-325. doi: 10.1016/j.xkme.2020.01.013. eCollection 2020 May-Jun. PMID 32734251